CLINICAL TRIAL: NCT02759185
Title: Placebo-Controlled, Triple-Blind, Randomized Crossover Pilot Study of the Safety and Efficacy of Four Different Potencies of Smoked Marijuana in 76 Veterans With Chronic, Treatment-Resistant Posttraumatic Stress Disorder (PTSD)
Brief Title: Pilot Study of the Safety and Efficacy of Four Different Potencies of Smoked Marijuana in 76 Veterans With PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MJP-1
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; marijuana; cannabis; sleep; THC; CBD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Marijuana Abuse | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High THC cannabis (Experimental): Provided up to 1.8 g of cannabis per day with more tetrahydrocannabinol than cannabidiol
  Interventions: Drug: High THC cannabis
- High CBD cannabis (Experimental): Provided up to 1.8 g of cannabis per day of marijuana with more cannabidiol than tetrahydrocannabinol
  Interventions: Drug: High CBD cannabis
- THC/CBD cannabis (Experimental): Provided up to 1.8 g of cannabis per day with an approximately equal amount of tetrahydrocannabinol and cannabidiol
  Interventions: Drug: THC/CBD cannabis
- Placebo cannabis (Placebo Comparator): Provided 1.8 g of cannabis per day with very low levels of tetrahydrocannabinol and cannabidiol
  Interventions: Drug: Placebo cannabis

INTERVENTIONS:
Drug: High THC cannabis — Three weeks of smoking cannabis containing more THC than CBD with amount smoked limited to no more than 1.8 g per day.
  Other Names: Tetrahydrocannabinol
  Arms: High THC cannabis
Drug: High CBD cannabis — Three weeks of smoking cannabis containing more CBD than THC with amount smoked limited to no more than 1.8 g per day.
  Other Names: Cannabidiol
  Arms: High CBD cannabis
Drug: THC/CBD cannabis — Three weeks of smoking cannabis containing equal amounts of THC and CBD with smoking limited to no more than 1.8 g per day.
  Other Names: Tetrahydrocannabinol; Cannabidiol
  Arms: THC/CBD cannabis
Drug: Placebo cannabis — Three weeks of smoking cannabis with low levels of THC and CBD with smoking limited to no more than 1.8 per day.
  Arms: Placebo cannabis

SUMMARY:
This pilot study gathered preliminary evidence of the safety and efficacy of four potencies of smoked cannabis to manage chronic, treatment-resistant PTSD among veterans: (1) High THC/ Low CBD (High THC), (2) Low THC/High CBD (High CBD), (3) High THC/ High CBD (THC/CBD) and (4) Low THC/Low CBD (placebo). The study will produce preliminary evidence to help elucidate the potential effects of THC, CBD, or a combination of both constituents to reduce PTSD symptoms. Smoked cannabis will be tested in two stages of three weeks each (Stage 1 and Stage 2), with a two-week cessation period after each stage, verified by blood/urine cannabinoid analysis. The primary objective was to compare three active concentrations of smoked cannabis and placebo on PTSD symptom severity measured by CAPS-5 total severity scores during Stage 1.

DETAILED DESCRIPTION:
PTSD is a serious, worldwide public health problem resulting from traumatic experiences such as sexual assault, war, or abuse. PTSD is associated with high rates of psychiatric and medical co-morbidity, disability, suffering, and suicide. Despite available treatments for PTSD, many individuals continue to experience marked PTSD symptoms following treatment. In response to overwhelming demand for new treatments, several U.S. states have passed laws allowing the medical use of cannabis by individuals with PTSD.

Emerging observational and early clinical evidence suggest that cannabis may have the potential to reduce or ameliorate a number of symptoms experienced by those with PTSD, including sleep difficulty and anxiety. Indeed, some evidence has suggested that delta-9-tetrahydrocannabinol (THC) may serve to reduce nightmares among those with PTSD, while other studies have shown anxiolytic effects of cannabidiol (CBD). However, there have been no randomized controlled trials of cannabis, in any form, for PTSD.

The present triple-blind, randomized, placebo-controlled crossover trial aims to examine the safety and efficacy of four types of cannabis (i.e., high THC, low CBD; high CBD, low THC; equal ratio THC/CBD; and placebo) among 76 military veterans with chronic treatment-resistant PTSD of at least six months' duration. The study will produce preliminary evidence to help elucidate the contribution of THC, CBD, or a combination of both constituents to potential attenuation of PTSD symptoms.

Smoked cannabis was tested in two stages lasting three weeks each (Stage 1 and Stage 2), with a two-week cessation after each stage, verified by blood/urine cannabinoid analysis. The primary objective was to compare three active concentrations of smoked cannabis and placebo on PTSD symptom severity measured by CAPS-5 total scores during Stage 1.

Study participants received one of four different types of cannabis during Stage 1 with crossover and re-randomization, less the placebo cannabis, at Stage 2. The four potencies of cannabis were High THC/ Low CBD (High THC), Low THC/High CBD (High CBD), High THC/High CBD (THC/CBD) and Low THC/Low CBD (placebo). "High" is defined as marijuana containing a target of 7-15% concentration by weight of the respective cannabinoid and "Low" is defined as < 2% concentration by weight. Prior to each stage, participants completed two introductory sessions where they were trained on cannabis self-administration. During each stage, participants were provided 1.8 grams of cannabis daily to smoke ad libitum. Each stage was followed by a two-week cessation period.

The primary objective was to compare three active concentrations of smoked cannabis and placebo on PTSD symptom severity measured by CAPS-5 total severity scores during Stage 1.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic treatment-resistant PTSD of at least six months duration.
* Have PTSD of at least moderate severity at the time of baseline assessment.
* Be a military veteran with PTSD.
* Be at least 18 years old.
* Be willing to commit to medication dosing and delivery method, to completing evaluation instruments, and attending all study visits.
* Agree to use only cannabis provided by site staff and agree to required cessation periods for the duration of the study.
* Report no current hazardous cannabis use and completely abstain from cannabis during the 2-week baseline assessment period (verified via urine and/or blood cannabinoid concentrations).
* Agree to video record all cannabis administrations and provide video to the site staff for review during study participation.
* Agree to keep all cannabis provided by site staff securely stored in the provided lock box and not to share/distribute cannabis to any other individual.
* Be stable on any pre-study medications and/or psychotherapy regimen for PTSD prior to study entry, agree to notify their physician/clinician about participation in the study, and agree to report any changes in medication or psychotherapy treatment regimen during the study, to site staff.
* If female and of childbearing potential, agree to use an effective form of birth control during study participation and may only be allowed to enroll and continue in the study based on a negative pregnancy test.
* Be proficient in reading and writing in English and able to effectively communicate with site staff.
* Agree not to participate in any other interventional clinical trials during the study

Exclusion Criteria:

* Upon review of medical or psychiatric history must not have any current or past diagnosis that would be considered a risk to participation in the study.
* Have any allergies to cannabis or contraindication for smoking of cannabis
* Are abusing illegal drugs.
* Are not able to give adequate informed consent.
* Are not able to attend face-to-face visits or those who plan to move out of the area within the treatment period.
* Are pregnant or nursing, or if a woman who can have children, those who are not practicing an effective means of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Sisley, MD, Principal Investigator — President of Scottsdale Research Institute
Locations (1):
- Scottsdale Research Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bonn-Miller MO, Sisley S, Riggs P, Yazar-Klosinski B, Wang JB, Loflin MJE, Shechet B, Hennigan C, Matthews R, Emerson A, Doblin R. The short-term impact of 3 smoked cannabis preparations versus placebo on PTSD symptoms: A randomized cross-over clinical trial. PLoS One. 2021 Mar 17;16(3):e0246990. doi: 10.1371/journal.pone.0246990. eCollection 2021. PMID 33730032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via letters of referral sent to psychiatrists and psychotherapists, contact with veterans' organizations, advertisements or announcements placed in appropriate locations or on appropriate internet sites and the sponsor site, and word of mouth.
Pre-assignment Details: For Stage 2, participants were re-randomized into one of three treatment groups which excluded placebo and their Stage 1 treatment assignment.
Groups:
- High THC Cannabis (Stage 1); High THC Cannabis (Stage 2): Provided up to 1.8 g of cannabis per day with more tetrahydrocannabinol than cannabidiol
  High THC cannabis: three weeks of smoked cannabis containing more THC than CBD, with amount smoked limited to no more than 1.8 g per day.
- High CBD Cannabis (Stage 1); High CBD Cannabis (Stage 2): Provided with up to 1.8 g of cannabis per day with more cannabidiol than tetrahydrocannabinol
  High CBD cannabis: three weeks of smoked cannabis containing more CBD than THC, with amount smoked limited to no more than 1.8 g per day.
- THC/CBD Cannabis (Stage 1); THC/CBD Cannabis (Stage 2): Provided up to 1.8 g of cannabis per day with an approximately equal amount of tetrahydrocannabinol and cannabidiol
  THC/CBD cannabis: three weeks of smoked cannabis containing equal amounts of THC and CBD, with amount smoked limited to no more than 1.8 g per day.
- Placebo Cannabis (Stage 1): Provided up to 1.8 g of cannabis per day with very low levels of tetrahydrocannabinol and cannabidiol
  Placebo cannabis: three weeks of smoked cannabis with low levels of THC and CBD, with amount smoked limited to no more than 1.8 per day.
Period: Stage 1
Arm/Group | High THC Cannabis (Stage 1) | High CBD Cannabis (Stage 1) | THC/CBD Cannabis (Stage 1) | Placebo Cannabis (Stage 1) | High THC Cannabis (Stage 2) | High CBD Cannabis (Stage 2) | THC/CBD Cannabis (Stage 2)
Started | 20 | 20 | 20 | 20 | 0 | 0 | 0
Completed | 19 | 19 | 17 | 20 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | High THC Cannabis (Stage 1) | High CBD Cannabis (Stage 1) | THC/CBD Cannabis (Stage 1) | Placebo Cannabis (Stage 1) | High THC Cannabis (Stage 2) | High CBD Cannabis (Stage 2) | THC/CBD Cannabis (Stage 2)
Started | 0 | 0 | 0 | 0 | 29 | 27 | 18
Completed | 0 | 0 | 0 | 0 | 27 | 24 | 17
Not Completed | 0 | 0 | 0 | 0 | 2 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) set
Groups:
- High THC Cannabis: Provided up to 1.8 g of cannabis per day with more tetrahydrocannabinol than cannabidiol
  High THC cannabis: Three weeks of smoking cannabis containing more THC than CBD, with amount smoked limited to no more than 1.8 g per day.
- High CBD Cannabis: Provided up to 1.8 g of cannabis per day of marijuana with more cannabidiol than tetrahydrocannabinol
  High CBD cannabis: Three weeks of smoking cannabis containing more CBD than THC, with amount smoked limited to no more than 1.8 g per day.
- High THC/ High CBD Cannabis: Provided up to 1.8 g of cannabis per day with an approximately equal amount of tetrahydrocannabinol and cannabidiol
  High THC/high CBD cannabis: Three weeks of smoking cannabis containing equal amounts of THC and CBD, with smoking limited to no more than 1.8 g per day.
- Placebo Cannabis: Provided 1.8 g of cannabis per day a with very low levels of tetrahydrocannabinol and cannabidiol
  Placebo cannabis: Three weeks of smoking cannabis with low levels of THC and CBD, with smoking limited to no more than 1.8 per day.
- Total: Total of all reporting groups
Arm/Group | High THC Cannabis | High CBD Cannabis | High THC/ High CBD Cannabis | Placebo Cannabis | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (16.6) | 40.4 (11.2) | 50.6 (13.3) | 43.7 (12.5) | 44.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 2 | 8
  Male | 19 | 18 | 17 | 18 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 11 | 14 | 14 | 14 | 53
  Race/Ethnicity: Other | 9 | 6 | 6 | 6 | 27
Education [Count of Participants; unit: Participants]
  High School Graduate | 0 | 3 | 1 | 2 | 6
  Some College/Associate's Degree | 13 | 10 | 8 | 11 | 42
  College Graduate | 7 | 7 | 11 | 7 | 32
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.0 (8.9) | 31.3 (6.6) | 31.4 (7.4) | 33.1 (7.0) | 31.9 (7.4)
Combat-related trauma (yes) [Count of Participants; unit: Participants] | 13 | 13 | 15 | 13 | 54
Sleep Apnea (STOP-bang) [Count of Participants; unit: Participants]
  Low risk = 1 | 6 | 6 | 4 | 6 | 22
  Intermediate risk = 2 | 3 | 3 | 3 | 3 | 12
  High risk = 3 | 11 | 11 | 13 | 11 | 46
Cannabis Use Disorders Identification Test-Revised (CUDIT-R) [Mean (Standard Deviation); unit: score on a scale] — The CUDIT-R is a brief cannabis screening tool to identify cannabis misuse. Participants who report past six month cannabis use are asked eight additional questions on cannabis where each item score range from 0 to 4. The total CUDIT-R score ranges from 0 to 24 with ≥ 8 indicating hazardous cannabis use and ≥ 12 indicating a possible cannabis use disorder.
  score on a scale | 3.9 (3.0) | 2.5 (2.8) | 2.4 (2.8) | 1.7 (2.6) | 2.6 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Baseline CAPS-5 Total Severity Score
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a CAPS-5 total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance), and D (hypervigilance), and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline (3 weeks after randomization)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High THC Cannabis: Provided up to 1.8 g of cannabis per day with more tetrahydrocannabinol than cannabidiol
  High THC cannabis: three weeks of smoked cannabis containing more THC than CBD, with amount smoked limited to no more than 1.8 g per day.
- High CBD Cannabis: Provided up to 1.8 g of cannabis per day where product has more cannabidiol than tetrahydrocannabinol
  High CBD cannabis: three weeks of smoked cannabis containing more CBD than THC, with amount smoked limited to no more than 1.8 g per day.
- THC/CBD Cannabis: Provided up to 1.8 g of cannabis per day with an approximately equal amount of tetrahydrocannabinol and cannabidiol
  THC/CBD cannabis: three weeks of smoked cannabis containing approximate equal amounts of THC and CBD, with amount smoked limited to no more than 1.8 g per day.
- Placebo Cannabis: Provided up to 1.8 g of cannabis per day with very low levels of tetrahydrocannabinol and cannabidiol
  Placebo cannabis: three weeks of smoked cannabis with low levels of THC and CBD, with amount smoked limited to no more than 1.8 per day.
Arm/Group | High THC Cannabis | High CBD Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 20 | 20 | 20 | 20
score on a scale | 36.6 (7.20) | 36.8 (8.23) | 38.0 (7.8) | 37.3 (6.38)

2. Primary Outcome: Stage 1 Primary Endpoint CAPS-5 Total Severity Scores (Visit 5)
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a CAPS-5 total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance), and D (hypervigilance); and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Visit 5 (between end of week 3 and start of week 4) of Stage 1
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High CBD Cannabis: Provided up to 1.8 g of cannabis per day with more cannabidiol than tetrahydrocannabinol
  High CBD cannabis: three weeks of smoked cannabis containing more CBD than THC, with amount smoked limited to no more than 1.8 g per day.
- THC/CBD Cannabis: Provided up to 1.8 g of cannabis per day with an approximately equal amount of tetrahydrocannabinol and cannabidiol
  High THC/high CBD cannabis: three weeks of smoked cannabis containing equal amounts of THC and CBD, with amount smoked limited to no more than 1.8 g per day.
- Placebo Cannabis: Provided with 1.8 g of cannabis per day with very low levels of tetrahydrocannabinol and cannabidiol
  Placebo cannabis: three weeks of smoked cannabis with low levels of THC and CBD, with amount smoked limited to no more than 1.8 per day.
Arm/Group | High THC Cannabis | High CBD Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 19 | 19 | 19 | 20
score on a scale | 20.5 (8.97) | 28.1 (13.26) | 29.6 (12.17) | 24.2 (12.79)

3. Primary Outcome: Change in CAPS-5 Total Severity Scores From Baseline to Stage 1 Primary Endpoint (Visit 5)
Description: as for outcome 2
Time Frame: Baseline (3 weeks after randomization) to Primary Endpoint (Visit 5, between end of week 3 and start of week 4)
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- THC/CBD Cannabis: Provided up to 1.8 g of cannabis per day with an approximately equal amount of tetrahydrocannabinol and cannabidiol
  THC/CBD cannabis: three weeks of smoked cannabis containing equal amounts of THC and CBD, with amount smoked limited to no more than 1.8 g per day.
Arm/Group | High THC Cannabis | High CBD Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 19 | 19 | 19 | 20
score on a scale | -15.2 (11.03) | -8.4 (10.09) | -8.5 (9.88) | -13.1 (12.10)

4. Secondary Outcome: Change in PTSD Checklist (PCL-5) From Baseline to Stage 1 Primary Endpoint
Description: The PTSD Checklist (PCL-5) is a 20-item self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms. Participants indicate how much distress they have experienced due to various PTSD symptoms on a five-point Likert-type scale (0=not at all, 4=extremely). The total PCL-5 score (a sum of all 20 items) ranges from 0 to 80, with higher scores indicating greater symptom severity.
Time Frame: Baseline (3 weeks after randomization) to Stage 1 Primary Endpoint (Visit 6, 3 weeks post self-administration and prior to cessation)
Population: Intent-to-treat (ITT) Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High THC Cannabis | High CBD Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 19 | 19 | 18 | 19
score on a scale | -23.5 (16.5) | -12.1 (16.2) | -16.4 (9.1) | -14.6 (15.6)

5. Secondary Outcome: Change in Inventory of Depression and Anxiety (IDAS) Social Anxiety Total Scores From Baseline to Stage 1 Primary Endpoint
Description: The Inventory of Depression and Anxiety (IDAS) is a 64-item self-report measure of non-overlapping scales that assess specific depression and anxiety symptoms. Respondents indicate on a scale of 1 (not at all) to 5 (extremely) how much they have felt or experienced several symptoms in the past two weeks. The IDAS consists of 10 symptom scales: Suicidality, Lassitude, Insomnia, Appetite Loss, Appetite Gain, Ill Temper, Well-Being, Panic, Social Anxiety, and Traumatic Intrusions. Items that assess social anxiety are summed and range from 5 to 25 with higher scores indicating greater anxiety symptoms.
Time Frame: as for outcome 4
Population: Intent-to-treat (ITT) set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High THC Cannabis | High CBD Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 19 | 19 | 18 | 19
score on a scale | -3.7 (4.2) | -2.7 (2.7) | -2.2 (2.0) | -2.4 (4.3)

6. Secondary Outcome: Change in Inventory of Psychosocial Functioning (IPF) From Baseline to Stage 1 Primary Endpoint
Description: The Inventory of Psychosocial Functioning (IPF) is an 80-item measure that was developed for use among individuals with PTSD. It assesses current psychosocial functioning across seven domains: romantic relationships, family, work, friendships, parenting, education, and self-care. Items are scored on a 0 (never) to 6 (always) scale. Summation of scores across domains yields a total score for psychosocial functioning, with higher scores indicating greater functional impairment.
Time Frame: as for outcome 4
Population: Intent-to-treat (ITT) Set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo Cannabis: Provided with 1.8 g of cannabis per day with very low levels of tetrahydrocannabinol and cannabidiol
  Placebo cannabis: three weeks of smoking cannabis with low levels of THC and CBD, with amount smoked limited to no more than 1.8 per day.
Arm/Group | High THC Cannabis | High CBD Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 19 | 19 | 18 | 20
score on a scale | 1.2 (11.9) | -1.2 (5.5) | 4.1 (8.5) | -0.2 (6.7)

7. Secondary Outcome: Change in Inventory of Depression and Anxiety (IDAS) General Depression Total Scores From Baseline to Stage 1 Primary Endpoint
Description: The Inventory of Depression and Anxiety (IDAS) is a 64-item self-report measure of non-overlapping scales that assess specific depression and anxiety symptoms. Respondents indicate on a scale of 1 (not at all) to 5 (extremely) how much they have felt or experienced several symptoms in the past two weeks. The IDAS consists of 10 symptom scales: Suicidality, Lassitude, Insomnia, Appetite Loss, Appetite Gain, Ill Temper, Well-Being, Panic, Social Anxiety, and Traumatic Intrusions. Items that assess general depression are summed and range from 20 to 100 with higher scores indicating greater depressive symptoms.
Time Frame: as for outcome 4
Population: Intent-to-treat (ITT) Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High THC Cannabis | High CBD Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 19 | 19 | 18 | 20
score on a scale | -16.1 (12.6) | -11.4 (11.7) | -13.4 (9.1) | -8.3 (11.2)

8. Secondary Outcome: Change in Insomnia Severity Index (ISI) Scores From Baseline to Stage 1 Primary Endpoint
Description: The Insomnia Severity Index (ISI) is a brief self-reported measure of insomnia. It consists of seven questions, with responses made on a five-point Likert scale. Three items address difficulty at sleep onset, maintaining sleep, and early waking, and four questions address perceived quality of sleep and effects of sleep difficulties on daily function. Questions are summed into a total score that ranges from 0 to 28 and can be interpreted as ranging from no signs of insomnia to severe insomnia. Higher scores indicate more severe insomnia.
Time Frame: as for outcome 4
Population: Intent-to-treat Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High THC Cannabis | High CBD Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 18 | 19 | 18 | 20
score on a scale | -8.8 (5.2) | -5.9 (6.5) | -6.6 (5.2) | -6.1 (5.7)

9. Other Pre Specified Outcome: Actigraph Change in Sleep Efficiency
Description: Daily sleep measures were collected using the Actigraph Watch at baseline and throughout the study period. Data were processed using the Actigraph Software according to the User Manual to measure "sleep efficiency," which is defined as the proportion of the estimated sleep periods spent asleep. Change in sleep efficiency was calculated and compared across the four treatment groups to assess whether there was any improvement or worsening in sleep efficiency before and after the 4-week treatment period. Other measures included number of days data were collected and average duration in minutes of time that were excluded and not recorded. Daily data were aggregated to analyze participants' average weekly sleep patterns.
Time Frame: Change in sleep efficiency from baseline to end of 4-week treatment period (visit 6)
Population: All participants were asked to wear the Actiwatch for sleep measures and all available data were analyzed to assess sleep efficiency. Note: the proportion of missing data prevented robust analysis and interpretation.
Measure: Mean (Standard Deviation); unit: percentage of total sleep time
Arm/Group | High CBD Cannabis | High THC Cannabis | THC/CBD Cannabis | Placebo Cannabis
Number analyzed (Participants) | 13 | 12 | 10 | 12
percentage of total sleep time | 0.17 (10.9) | 6.83 (6.55) | 1.80 (8.39) | -0.28 (6.36)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (Approximately 8 months)
Groups:
- High CBD Cannabis (Stage 1); High CBD Cannabis (Stage 2): Provided up to 1.8 g of cannabis per day with more cannabidiol than tetrahydrocannabinol
  High CBD cannabis: three weeks of smoked cannabis containing more CBD than THC, with amount smoked limited to no more than 1.8 g per day.
- Placebo Cannabis (Stage 1): Provided with 1.8 g of cannabis per day with very low levels of tetrahydrocannabinol and cannabidiol
  Placebo cannabis: three weeks of smoked cannabis with low levels of THC and CBD, with amount smoked limited to no more than 1.8 per day.
- THC/CBD Cannabis (Stage 2): Provided up to 1.8 g of cannabis per day with an approximately equal amount of tetrahydrocannabinol and cannabidiol
  THC/CBD cannabis: three weeks of smoked cannabis containing more CBD than THC, with amount smoked limited to no more than 1.8 g per day.
Arm/Group | High THC Cannabis (Stage 1) | High CBD Cannabis (Stage 1) | THC/CBD Cannabis (Stage 1) | Placebo Cannabis (Stage 1) | High THC Cannabis (Stage 2) | High CBD Cannabis (Stage 2) | THC/CBD Cannabis (Stage 2)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/29 | 0/27 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 3/20 | 0/20 | 1/29 | 1/27 | 0/18
Other Adverse Events (participants affected / at risk) | 17/20 | 19/20 | 19/20 | 18/20 | 22/29 | 22/27 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High THC Cannabis (Stage 1) (N=20) | High CBD Cannabis (Stage 1) (N=20) | THC/CBD Cannabis (Stage 1) (N=20) | Placebo Cannabis (Stage 1) (N=20) | High THC Cannabis (Stage 2) (N=29) | High CBD Cannabis (Stage 2) (N=27) | THC/CBD Cannabis (Stage 2) (N=18)
Heart palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High THC Cannabis (Stage 1) (N=20) | High CBD Cannabis (Stage 1) (N=20) | THC/CBD Cannabis (Stage 1) (N=20) | Placebo Cannabis (Stage 1) (N=20) | High THC Cannabis (Stage 2) (N=29) | High CBD Cannabis (Stage 2) (N=27) | THC/CBD Cannabis (Stage 2) (N=18)
Dry eye (Eye disorders) | 3 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 5 | 1 | 3 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1 | 2 | 5 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 2 | 2 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 2 | 0 | 2 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 4 | 5 | 2 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 0 | 0 | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 5 | 2 | 2 | 3 | 6 | 4 | 1
Depression (Psychiatric disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 1
Irritability (Psychiatric disorders) | 3 | 0 | 1 | 0 | 1 | 3 | 3
Libido increased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Paranoia (Psychiatric disorders) | 3 | 0 | 3 | 0 | 3 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2 | 2 | 2 | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 6 | 2 | 1 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth repair (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anger (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hostility (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Wisdom teeth removal (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal infections (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Obsessive thoughts (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicide ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT02759185/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT02759185/SAP_001.pdf
  • Informed Consent Form (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT02759185/ICF_002.pdf